CLINICAL TRIAL: NCT02446600
Title: A Phase III Study Comparing Single-Agent Olaparib or the Combination of Cediranib and Olaparib to Standard Platinum-Based Chemotherapy in Women With Recurrent Platinum-Sensitive Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Testing the Use of A Single Drug (Olaparib) or the Combination of Two Drugs (Cediranib and Olaparib) Compared to the Usual Chemotherapy for Women With Platinum Sensitive Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: AstraZeneca (Industry); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00606; NCI-2015-00606 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s16-01480; NRG-GY004; NRG-GY004 (Other: NRG Oncology); NRG-GY004 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2015-05-11; First posted 2015-05-18 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-08

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Tumor; Ovarian Seromucinous Carcinoma; Ovarian Serous Tumor; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Ovarian Endometrioid Adenocarcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Specimen Handling; Carboplatin; cediranib; Gemcitabine; Magnetic Resonance Spectroscopy; olaparib; Paclitaxel; Taxes; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (platinum-based chemotherapy) (Active Comparator): See detailed description.
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Gemcitabine; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Other: Quality-of-Life Assessment
- Arm II (olaparib) (Experimental): Patients receive olaparib PO BID. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening. Patients also undergo CT or MRI as well as blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Olaparib; Other: Pharmacological Study; Other: Quality-of-Life Assessment
- Arm III (olaparib, cediranib maleate) (Experimental): Patients receive olaparib PO BID and cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo CT or MRI as well as blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Olaparib; Other: Pharmacological Study; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm II (olaparib); Arm III (olaparib, cediranib maleate)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (platinum-based chemotherapy)
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
  Arms: Arm III (olaparib, cediranib maleate)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
  Arms: Arm I (platinum-based chemotherapy)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
  Arms: Arm I (platinum-based chemotherapy)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Arm II (olaparib); Arm III (olaparib, cediranib maleate)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (platinum-based chemotherapy)
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
  Arms: Arm I (platinum-based chemotherapy)
Other: Pharmacological Study — Correlative studies
  Arms: Arm II (olaparib); Arm III (olaparib, cediranib maleate)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase III trial studies olaparib or cediranib maleate and olaparib to see how well they work compared with standard platinum-based chemotherapy in treating patients with platinum-sensitive ovarian, fallopian tube, or primary peritoneal cancer that has come back. Olaparib and cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Cediranib maleate may stop the growth of ovarian, fallopian tube, or primary peritoneal cancer by blocking the growth of new blood vessels necessary for tumor growth. Drugs used in chemotherapy, such as carboplatin, paclitaxel, gemcitabine hydrochloride, and pegylated liposomal doxorubicin hydrochloride work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether olaparib or cediranib maleate and olaparib is more effective than standard platinum-based chemotherapy in treating patients with platinum-sensitive ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the efficacy of either single agent olaparib or the combination of cediranib (cediranib maleate) and olaparib, as measured by progression free survival (PFS), as compared to standard platinum-based chemotherapy in the setting of recurrent platinum-sensitive ovarian, primary peritoneal or fallopian tube cancer.

SECONDARY OBJECTIVES:

I. Assess the efficacy of single agent olaparib or the combination of cediranib and olaparib, as measured by response rate and overall survival as compared to standard platinum-based chemotherapy in the setting of recurrent platinum-sensitive ovarian, primary peritoneal or fallopian tube cancer.

II. Assess the efficacy of single agent olaparib or the combination of cediranib and olaparib, as measured by PFS, in women with or without deleterious germline breast cancer (BRCA) mutations (gBRCAmt) in the setting of recurrent platinum-sensitive ovarian, primary peritoneal, or fallopian tube cancer.

III. Assess the effect on disease-related symptoms (DRS) as measured by the 9-item DRS-P subscale of the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy (NCCN-FACT) Ovarian Symptom Index-18 (NFOSI-18), of single agent olaparib or cediranib and olaparib, compared to standard platinum-based chemotherapy, in the setting of recurrent platinum sensitive ovarian, primary peritoneal or fallopian tube cancer.

IV. Assess the efficacy of single agent olaparib or the combination of cediranib and olaparib, as measured by PFS, in women with or without homologous repair deficiencies as measured by BROCA in the setting of recurrent platinum-sensitive ovarian, primary peritoneal, or fallopian tube cancer.

V. To assess changes in the number of circulating endothelial cells (CECs) following three days of treatment with olaparib, combination olaparib/cediranib, or standard platinum-based chemotherapy in women with recurrent platinum-sensitive ovarian, primary peritoneal, or fallopian tube cancer.

VI. To assess whether change in the number of circulating endothelial cells (CECs) following three days of treatment with olaparib, combination olaparib/cediranib, or standard platinum-based chemotherapy in women with recurrent platinum-sensitive ovarian, primary peritoneal, or fallopian tube cancer is prognostic for PFS.

VII. To develop a profile from a panel of angiogenic biomarkers in women with recurrent platinum-sensitive ovarian, primary peritoneal, or fallopian tube cancer which is associated with PFS, and then validate the predictive value of this biomarker profile.

EXPLORATORY OBJECTIVES:

I. To assess the time from randomization to the first non-study, anti-cancer therapy, surgery or death (TFST) for single-agent olaparib or combination cediranib and olaparib relative to standard platinum-based chemotherapy in the setting of recurrent platinum-sensitive ovarian, primary peritoneal or fallopian tube cancer.

II. To assess the time from randomization to the second non-study, anti-cancer therapy, surgery or death (TSST) for single-agent olaparib or combination cediranib and olaparib relative to standard platinum-based chemotherapy in the setting of recurrent platinum-sensitive ovarian, primary peritoneal or fallopian tube cancer.

III. Assess the effect on secondary measures of quality of life, as assessed by the treatment side effects (TSE) and function/well-being (F/WB) subscales of the NFOSI-18, sensory neuropathy as measured by the FACT/Gynecologic Oncology Group-Neurotoxicity version 4 (GOG-Ntx-4), and health utility as measured by the Euro Quality of Life-5 Dimension (EQ-5D), of single agent olaparib or cediranib and olaparib, compared to standard platinum-based chemotherapy, in the setting of recurrent platinum sensitive ovarian, primary peritoneal or fallopian tube cancer.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients may be treated with one of the three regimens per investigator discretion.

REGIMEN I: Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30-60 minutes and on day 1. Treatment repeats every 21 days for at least 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) as well as blood sample collection throughout the trial.

REGIMEN II: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 for at least 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening. Patients also undergo CT or MRI as well as blood sample collection throughout the trial.

REGIMEN III: Patients receive pegylated liposomal doxorubicin hydrochloride IV and carboplatin IV over 30-60 minutes and on day 1. Treatment repeats every 28 days for at least 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo CT or MRI as well as blood sample collection throughout the trial.

ARM II: Patients receive olaparib orally (PO) twice daily (BID). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening. Patients also undergo CT or MRI as well as blood sample collection throughout the trial.

ARM III: Patients receive olaparib PO BID and cediranib maleate PO once daily (QD). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo CT or MRI as well as blood sample collection throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have platinum-sensitive recurrent high-grade serous or high-grade endometrioid ovarian, primary peritoneal, or fallopian tube cancers; patients with other (clear cell, mixed epithelial, undifferentiated carcinoma, or transitional cell carcinoma) high-risk histologies are also eligible, provided that the patient has a known deleterious germline BRCA1 or BRCA2 mutation identified through testing at a clinical laboratory; Note: Due to the long acceptance of germline BRCA testing through Myriad, Myriad testing will be accepted; if testing for germline BRCA is done by other organizations, documentation from a qualified medical professional (e.g., ovarian cancer specialty physician involved in the field, high risk genetics physician, genetics counselor) listing the mutation and confirming that the laboratory results showed a recognized germline deleterious BRCA1 or BRCA2 mutation or BRCA rearrangement is required; please collect a copy of Myriad or other BRCA mutational analysis (positive or VUS or negative) reports

  * Platinum-sensitive disease defined as no clinical or radiographic evidence of disease recurrence for > 6 months (or 182 days) after last receipt of platinum-based therapy
  * Patients must have had a complete clinical response to their prior line of platinum therapy and cannot have had progression through prior platinum-based therapy
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must have evaluable disease - defined as one of the following:

  * Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 measurable disease OR
  * Evaluable disease (defined as solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions OR ascites and/or pleural effusion that has been pathologically demonstrated to be disease-related) AND a cancer antigen 125 (CA125) that has doubled from the post-treatment nadir and is also greater than 2 times upper limit of normal (ULN)
* Prior therapy:

  * Prior chemotherapy must have included a first-line platinum-based regimen with or without intravenous consolidation chemotherapy
  * Patients may have received an unlimited number of platinum-based therapies in the recurrent setting
  * Patients may have received up to 1 non-platinum-based line of therapy in the recurrent setting; prior hormonal therapy will not be considered to count as this non-platinum-based line
  * Patients may not have had a prior anti-angiogenic agent in the recurrent setting; prior use of bevacizumab in the upfront or upfront maintenance setting is allowed
  * Patients may not have previously received a poly adenosine diphosphate (ADP) ribose polymerase (PARP)-inhibitor
  * Prior hormonal-based therapy for ovarian, primary peritoneal, or fallopian tube cancer is acceptable
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 10 g/dL
* Creatinine =< the institutional upper limit of normal (ULN) OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Urine protein: creatinine ratio (UPC) of =< 1 or less than or equal to 2+ proteinuria on two consecutive dipsticks taken no less than 1 week apart; UPC is the preferred test; patients with >= 2+ proteinuria on dipstick must also have a 24 hour urine collection demonstrating =< 500 mg over 24 hours
* Total bilirubin =< 1.5 x the institutional ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 times institutional ULN
* Toxicities of prior therapy (excepting alopecia) should be resolved to less than or equal to grade 1 as per National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE); patients with long-standing stable grade 2 neuropathy may be considered after discussion with the overall principal investigator (PI), but may not receive carboplatin and paclitaxel as the reference regimen, if randomized to that arm
* Patients must be able to swallow and retain oral medications and without gastrointestinal illnesses that would preclude absorption of cediranib or olaparib
* Patients must have adequately controlled blood pressure (BP), with a BP no greater than 140 mmHg (systolic) and 90 mmHg (diastolic) for eligibility; patients must have a BP of =< 140/90 mmHg taken in the clinic setting by a medical professional within 2 weeks prior to starting study; patients with hypertension may be managed with up to a maximum of three antihypertensive medications; it is strongly recommended that patients who are on three antihypertensive medications be followed by a cardiologist or blood pressure specialist for management of blood pressure while on protocol
* Patients must be willing and able to check and record daily blood pressure readings; blood pressure cuffs will be provided to patients randomized to Arm III
* Cediranib has been shown to terminate fetal development in the rat, as expected for a process dependent on VEGF signaling; for this reason, women of child-bearing potential must have a negative pregnancy test prior to study entry; women of child-bearing potential must agree to use two reliable forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 weeks after cediranib discontinuation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Adequately controlled thyroid function, with no symptoms of thyroid dysfunction and thyroid stimulating hormone (TSH) within normal limits
* Age >= 18

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) of starting treatment or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; patients may not have had hormonal therapy within 2 weeks prior to entering the study; patients receiving raloxifene for bone health as per Food and Drug Administration (FDA) indication may remain on raloxifene absent other drug interactions
* Patients may not be receiving any other investigational agents nor have participated in an investigational trial within the past 4 weeks
* Patients may not be receiving any medication that may markedly affect renal function (e.g., vancomycin, amphotericin, pentamidine)
* Patients may not have received prior treatment affecting the vascular endothelial growth factor (VEGF) pathway (including, but not limited to thalidomide, sunitinib, pazopanib, sorafenib, and nintedanib); bevacizumab used in the upfront setting in conjunction with chemotherapy and/or as maintenance to treat newly diagnosed disease will be allowed
* Patients may not have previously received a PARP inhibitor
* CA-125 only disease without RECIST 1.1 measurable or otherwise evaluable disease
* Patients with untreated brain metastases, spinal cord compression, or evidence of symptomatic brain metastases or leptomeningeal disease as noted on CT or MRI scans should not be included on this study, since neurologic dysfunction may confound the evaluation of neurologic and other adverse events; screening imaging to rule out brain metastases is not required for screening, but should be performed prior to study enrollment if clinically indicated; patients with treated brain metastases and resolution of any associated symptoms must demonstrate stable post-therapeutic imaging for at least 6 months following therapy prior to starting study drug
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cediranib or olaparib
* Participants receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) are ineligible; strong inhibitors and inducers of UGT/PgP should be used with caution
* History of gastrointestinal perforation; patients with a history of abdominal fistula will be considered eligible if the fistula was surgically repaired or has healed, there has been no evidence of fistula for at least 6 months, and patient is deemed to be at low risk of recurrent fistula
* History of intra-abdominal abscess within the past 3 months
* Current signs and/or symptoms of bowel obstruction or signs and/or symptoms of bowel obstruction within 3 months prior to starting study drugs
* Dependency on intravenous (IV) hydration or total parenteral nutrition (TPN)
* Any concomitant or prior invasive malignancies with the following curatively treated exceptions:

  * Treated limited stage basal cell or squamous cell carcinoma of the skin
  * Carcinoma in situ of the breast or cervix
  * Primary endometrial cancer meeting the following conditions: stage not greater than IA, grade 1 or 2, no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous/serous, clear cell, or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
  * Prior cancer treated with a curative intent with no evidence of recurrent disease 3 years following diagnosis and judged by the investigator to be at low risk of recurrence
* Patients with any of the following:

  * History of myocardial infarction within six months
  * Unstable angina
  * Resting electrocardiogram (ECG) with clinically significant abnormal findings
  * New York Heart Association (NYHA) classification of III or IV
* If cardiac function assessment is clinically indicated or performed: left ventricular ejection fraction (LVEF) less than normal per institutional guidelines, or < 55%, if threshold for normal not otherwise specified by institutional guidelines

  * Patients with the following risk factors should have a baseline cardiac function assessment:

    * Prior treatment with anthracyclines
    * Prior treatment with trastuzumab
    * Prior central thoracic radiation therapy (RT), including RT to the heart
    * History of myocardial infarction within 6 to 12 months (patients with history of myocardial infarction within 6 months are excluded from the study)
    * Prior history of impaired cardiac function
* History of stroke or transient ischemic attack within six months
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Clinically significant peripheral vascular disease or vascular disease (including aortic aneurysm or aortic dissection)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting cediranib
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (other than atrial fibrillation with controlled ventricular rate), or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because cediranib and olaparib are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with cediranib and olaparib, breastfeeding should be discontinued if the mother is treated with cediranib or olaparib; these potential risks may also apply to other agents used in this study
* Known HIV-positive individuals are ineligible because of the potential for pharmacokinetic interactions with cediranib or olaparib; in addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Patients may not use any complementary or alternative medicines including natural herbal products or folk remedies as they may interfere with the effectiveness of the study treatments
* No features suggestive of myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML) on peripheral blood smear or bone marrow biopsy, if clinically indicated
* No prior allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUBCT)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2020-02-23 (Actual); Study Completion 2026-08-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce F Liu, Principal Investigator — NRG Oncology
Locations (356):
- United States (337):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - Arizona Oncology Associates-Wilmot, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Marin Cancer Care Inc, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Women's Cancer Care-Covington, Covington, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Green Bay Oncology-Manistique, Manistique, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Texas Oncology-The Woodlands, The Woodlands, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - Women's Cancer Center of Seattle, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Canada (13):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
- Japan (5):
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - The Cancer Institute Hospital Of JFCR, Koto-ku, Tokyo
  - Saitama Medical University International Medical Center, Saitama
  - National Cancer Center Hospital, Tokyo
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Liu JF, Brady MF, Matulonis UA, Miller A, Kohn EC, Swisher EM, Cella D, Tew WP, Cloven NG, Muller CY, Bender DP, Moore RG, Michelin DP, Waggoner SE, Geller MA, Fujiwara K, D'Andre SD, Carney M, Alvarez Secord A, Moxley KM, Bookman MA. Olaparib With or Without Cediranib Versus Platinum-Based Chemotherapy in Recurrent Platinum-Sensitive Ovarian Cancer (NRG-GY004): A Randomized, Open-Label, Phase III Trial. J Clin Oncol. 2022 Jul 1;40(19):2138-2147. doi: 10.1200/JCO.21.02011. Epub 2022 Mar 15. PMID 35290101
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened for accrual February 4th, 2016. Accrual to the randomized component of this study stopped on November 13, 2017 after enrolling 579 patients. One enrollment was a duplicate, so data is reported for 578 subjects.
Groups:
- Arm I (Platinum-based Chemotherapy): REGIMEN I: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for at least 4 cycles in the absence of disease progression or unacceptable toxicity.
- Arm II (Olaparib): Patients receive olaparib PO BID. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm III (Olaparib, Cediranib Maleate): Patients receive olaparib PO BID and cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Japanese Cohort: A small Japanese run-in cohort to assess the toxicity profile and the frequency of unexpected toxicities in the Japanese population when the olaparib and cediranib combination is administered
Period: Overall Study
Arm/Group | Arm I (Platinum-based Chemotherapy) | Arm II (Olaparib) | Arm III (Olaparib, Cediranib Maleate) | Japanese Cohort
Started | 187 | 190 (Duplicate enrollment patient has been excluded from all analyses.) | 189 | 13
Completed | 147 (Completed status includes all clinical reasons for suspending treatment, including disease progression, death and adverse events.) | 178 (Completed status includes all clinical reasons for suspending treatment, including disease progression, death and adverse events.) | 162 (Completed status includes all clinical reasons for suspending treatment, including disease progression, death and adverse events.) | 12 (Completed status includes all clinical reasons for suspending treatment, including disease progression, death and adverse events.)
Not Completed | 40 | 12 | 27 | 1
Not completed — Never treated | 20 | 2 | 6 | 0
Not completed — Withdrawal by Subject | 19 | 5 | 17 | 0
Not completed — Ineligible | 1 | 4 | 4 | 1
Not completed — Duplicate Enrollment | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and Treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Platinum-based Chemotherapy) | Arm II (Olaparib) | Arm III (Olaparib, Cediranib Maleate) | Japanese Cohort | Total
Number analyzed (Participants) | 187 | 189 | 189 | 13 | 578
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.0) | 64.6 (10.0) | 64.0 (9.8) | 58.6 (8.3) | 62.6 (9.5)
Age, Customized [Count of Participants; unit: Participants]
  Less than 40 years | 4 | 3 | 1 | 0 | 8
  40-49 years | 10 | 11 | 13 | 2 | 36
  50-59 years | 53 | 48 | 52 | 5 | 158
  60-69 years | 74 | 63 | 71 | 5 | 213
  >= 70 years | 46 | 64 | 52 | 1 | 163
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 189 | 189 | 13 | 578
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 2 | 6 | 0 | 18
  Not Hispanic or Latino | 171 | 184 | 177 | 13 | 545
  Unknown or Not Reported | 6 | 3 | 6 | 0 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4 | 0 | 8
  Asian | 5 | 8 | 6 | 13 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 4 | 0 | 0 | 4
  Black or African American | 6 | 7 | 8 | 0 | 21
  White | 164 | 161 | 163 | 0 | 488
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 8 | 8 | 8 | 0 | 24

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Determined Using Response Evaluation Criteria in Solid Tumors Version 1.1 Criteria
Description: Progression free survival (PFS) was defined as the number of months between study enrollment and documentation of disease progression (RECIST 1.1) or death from any cause. Patients still alive and disease free at the last follow-up were censored on the date of last CT Scan, or the CT Scan date prior to two missed assessments. Japanese cohort not included in progression free survival analysis, only included in toxicity assessments.
Time Frame: The protocol required lesion assessments every 9 weeks from cycle 1, day 1 for the first year, then every 12 weeks thereafter until disease progression. An average of approximately 10 months.
Population: All Randomized subjects
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Platinum-based Chemotherapy) | Arm II (Olaparib) | Arm III (Olaparib, Cediranib Maleate)
Number analyzed (Participants) | 187 | 189 | 189
months | 10.3 [8.7 to 11.2] | 8.2 [6.6 to 8.7] | 10.4 [8.5 to 12.5]
Statistical Analysis 1: Comparison: Arm I (Platinum-based Chemotherapy) vs Arm III (Olaparib, Cediranib Maleate); Arm II was suspended for futility at the interim analysis so was not analyzed at the final analysis; Test type: Superiority; p = 0.077, Log Rank — The p-value is one-sided. Per the protocol, the statistical significance threshold was <0.025. Type 1 error was controlled using hierarchical testing strategy; The log rank test was stratified by the minimization factors provided at randomization; Hazard Ratio (HR) = 0.856, 95% CI 2-sided [0.663 to 1.105] — The hazard ratio estimate compares olaparib+cedirinib to chemotherapy. If olaparib+cedirinib is superior, the hazard ratio is <1.0

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the number of months between study enrollment and death from any cause. Patients still alive at the last follow-up were censored on the date of last contact. Japanese cohort not included in overall survival analysis, the cohort was only included in toxicity assessments.
Time Frame: Approximately 30 months
Population: All randomized subjects
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Platinum-based Chemotherapy) | Arm II (Olaparib) | Arm III (Olaparib, Cediranib Maleate)
Number analyzed (Participants) | 187 | 189 | 189
months | 31.3 [26.4 to 34.4] | 29.2 [23.9 to 32.7] | 30.5 [27.0 to 36.5]

3. Secondary Outcome: Frequency and Severity of Adverse Effects
Description: Number of treated patients with Adverse Events (grade 3 or higher) observed while receiving randomized therapy, by Preferred term with incidence rate greater than 5%.
Time Frame: During treatment period and up to 100 days after stopping the study treatment, up to 39 months.
Population: Treated with randomized therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Platinum-based Chemotherapy) | Arm II (Olaparib) | Arm III (Olaparib, Cediranib Maleate) | Japanese Cohort
Number analyzed (Participants) | 171 | 188 | 188 | 13
Participants
  Anemia | 23 | 28 | 11 | 1
  Fatigue | 3 | 12 | 31 | 0
  Neutrophil count decreased | 51 | 3 | 7 | 1
  Platelet count decreased | 24 | 2 | 3 | 0
  Urinary tract infection | 10 | 11 | 15 | 0
  White blood cell decreased | 22 | 3 | 2 | 1

4. Secondary Outcome: Patient Reported Scores of Disease-related Symptoms as Measured by the National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Ovarian Symptom Index-18 Disease-Related Symptom-Physical
Description: Disease-related physical symptoms were measured by the Disease-Related Symptom-Physical (DRS-P) subscale of the National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Ovarian Symptom Index-18 (NCCN/FOSI-18). The DRS-P subscale is composed of 9 items. For the negative statements (or questions), reversal was performed prior to score calculation. According to the FACIT measurement system, a subscale score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the subscale. The DRS-P score ranges 0-36 with a larger score suggesting better QOL (Quality of Life) or less symptoms. This analysis did not include the Japanese cohort.
Time Frame: Prior to cycle 1, week 12, week 24, week 36, week 48, week 60, week 72, week 84, week 96 and 108 weeks after starting treatment
Population: Subjects who have completed baseline and at least one follow-up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Platinum-based Chemotherapy) | Arm II (Olaparib) | Arm III (Olaparib, Cediranib Maleate)
Number analyzed (Participants) | 151 | 171 | 167
score on a scale
  Baseline | 17.1 (3.0) | 17.8 (2.7) | 17.9 (2.5)
  12 Weeks | 16.5 (2.8) | 17.4 (2.4) | 15.9 (3.0)
  24 Weeks | 16.3 (3.0) | 17.4 (2.8) | 16.3 (2.9)
  36 Weeks | 16.9 (3.0) | 17.2 (3.0) | 16.3 (2.7)
  48 Weeks | 16.9 (3.9) | 17.1 (2.6) | 16.5 (2.7)
  60 Weeks | 16.5 (3.6) | 16.9 (3.0) | 16.3 (2.7)
  72 Weeks | 17.1 (2.9) | 17.3 (2.7) | 16.3 (3.2)
  84 Weeks | 17.4 (2.9) | 17.2 (2.8) | 16.6 (2.7)
  96 Weeks | 17.0 (3.0) | 16.9 (2.6) | 17.0 (2.9)
  108 Weeks | 17.3 (2.5) | 17.4 (2.3) | 17.2 (2.4)

5. Other Pre Specified Outcome: Time From Randomization to the First Non-study, Anti-cancer Treatment or Death
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Time From Randomization to the Second Non-study, Anti-cancer Treatment or Death
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Starting with the first treatment received, and ending 100 days after the last treatment, or at the last following, whichever is sooner, up to 39 months.
Description: Eligible and treated participants were affected if they experienced grade 1-5 adverse event
Arm/Group | Arm I (Platinum-based Chemotherapy) | Arm II (Olaparib) | Arm III (Olaparib, Cediranib Maleate) | Japanese Cohort
All-Cause Mortality (participants affected / at risk) | 72/187 | 95/189 | 84/189 | 4/13
Serious Adverse Events (participants affected / at risk) | 18/187 | 22/189 | 29/189 | 1/13
Other Adverse Events (participants affected / at risk) | 169/187 | 184/189 | 184/189 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Platinum-based Chemotherapy) (N=187) | Arm II (Olaparib) (N=189) | Arm III (Olaparib, Cediranib Maleate) (N=189) | Japanese Cohort (N=13)
Anemia (Blood and lymphatic system disorders) | 2 | 9 | 4 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0
Asystole (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Chest Pain - Cardiac (Cardiac disorders) | 0 | 1 | 0 | 0
Eye Disorders - Other (Eye disorders) | 1 | 0 | 0 | 0
Duodenal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colonic Obstruction (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Colonic Perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 0
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 3 | 6 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Edema Limbs (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 2 | 0
Death Nos (General disorders) | 1 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 2 | 0
Infusion Related Reaction (General disorders) | 1 | 0 | 0 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Infections And Infestations - Other (Infections and infestations) | 0 | 0 | 1 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 2 | 0
Pelvic Infection (Infections and infestations) | 0 | 1 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 3 | 0
Enterocolitis Infectious (Infections and infestations) | 2 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 3 | 0 | 0 | 0
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 0 | 1 | 0 | 0
Creatinine Increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil Count Decreased (Investigations) | 2 | 1 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Musculoskeletal And Connective Tissue Disorder - O (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Treatment Related Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Stroke (Nervous system disorders) | 1 | 0 | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial Hemorrhage (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 0 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0
Thromboembolic Event (Vascular disorders) | 1 | 1 | 1 | 0
Peripheral Ischemia (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 12 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Platinum-based Chemotherapy) (N=187) | Arm II (Olaparib) (N=189) | Arm III (Olaparib, Cediranib Maleate) (N=189) | Japanese Cohort (N=13)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Hemolytic Uremic Syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 | 6 | 9 | 0
Anemia (Blood and lymphatic system disorders) | 96 | 94 | 37 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 2 | 2 | 0
Asystole (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 4 | 0
Palpitations (Cardiac disorders) | 7 | 2 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Heart Failure (Cardiac disorders) | 1 | 0 | 0 | 0
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 1 | 1 | 1 | 0
Cardiac Disorders - Other (Cardiac disorders) | 0 | 0 | 3 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 6 | 1 | 5 | 0
Chest Pain - Cardiac (Cardiac disorders) | 0 | 2 | 4 | 0
Middle Ear Inflammation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ear And Labyrinth Disorders - Other (Ear and labyrinth disorders) | 1 | 1 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 4 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 8 | 8 | 8 | 0
Hearing Impaired (Ear and labyrinth disorders) | 3 | 2 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 3 | 2 | 8 | 0
Hypothyroidism (Endocrine disorders) | 3 | 4 | 60 | 7
Hyperthyroidism (Endocrine disorders) | 3 | 2 | 14 | 0
Endocrine Disorders - Other (Endocrine disorders) | 0 | 0 | 6 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 1 | 1
Eye Disorders - Other (Eye disorders) | 4 | 1 | 6 | 0
Watering Eyes (Eye disorders) | 0 | 3 | 2 | 0
Eye Pain (Eye disorders) | 2 | 1 | 2 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 2 | 1 | 3 | 0
Photophobia (Eye disorders) | 1 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Blurred Vision (Eye disorders) | 16 | 6 | 15 | 0
Dry Eye (Eye disorders) | 1 | 0 | 3 | 0
Retinal Detachment (Eye disorders) | 0 | 1 | 0 | 0
Floaters (Eye disorders) | 0 | 2 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 3 | 7 | 0
Dyspepsia (Gastrointestinal disorders) | 14 | 26 | 18 | 0
Duodenal Obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Duodenal Fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 4 | 6 | 25 | 0
Colonic Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colonic Obstruction (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Colonic Perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colonic Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 6 | 0
Constipation (Gastrointestinal disorders) | 71 | 70 | 61 | 1
Diarrhea (Gastrointestinal disorders) | 40 | 51 | 151 | 11
Vomiting (Gastrointestinal disorders) | 39 | 65 | 84 | 6
Bloating (Gastrointestinal disorders) | 7 | 23 | 17 | 0
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomach Pain (Gastrointestinal disorders) | 3 | 2 | 6 | 1
Salivary Duct Inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 | 8 | 9 | 1
Anal Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Rectal Mucositis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 38 | 60 | 78 | 1
Periodontal Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 3 | 4 | 0
Oral Dysesthesia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Mucositis Oral (Gastrointestinal disorders) | 43 | 20 | 64 | 4
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 | 12 | 11 | 0
Anal Pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Oral Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Ileus (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Ileal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oral Pain (Gastrointestinal disorders) | 3 | 6 | 11 | 0
Abdominal Distension (Gastrointestinal disorders) | 4 | 9 | 11 | 1
Nausea (Gastrointestinal disorders) | 108 | 120 | 135 | 7
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 12 | 10 | 15 | 0
Rectal Pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Gastric Perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Jejunal Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Fecal Incontinence (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1 | 3 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 4 | 2 | 4 | 0
Ascites (Gastrointestinal disorders) | 1 | 9 | 5 | 2
Toothache (Gastrointestinal disorders) | 2 | 0 | 6 | 0
Esophageal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Flatulence (Gastrointestinal disorders) | 2 | 7 | 9 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
General Disorders And Administration Site Conditio (General disorders) | 3 | 5 | 8 | 0
Pain (General disorders) | 15 | 18 | 25 | 0
Neck Edema (General disorders) | 1 | 1 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 3 | 2 | 4 | 7
Localized Edema (General disorders) | 1 | 6 | 0 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0
Flu Like Symptoms (General disorders) | 14 | 5 | 6 | 0
Non-Cardiac Chest Pain (General disorders) | 3 | 4 | 12 | 0
Edema Limbs (General disorders) | 16 | 31 | 24 | 2
Edema Face (General disorders) | 3 | 0 | 2 | 1
Fatigue (General disorders) | 104 | 125 | 148 | 2
Death Nos (General disorders) | 1 | 1 | 0 | 0
Fever (General disorders) | 12 | 17 | 9 | 1
Gait Disturbance (General disorders) | 3 | 4 | 1 | 0
Chills (General disorders) | 10 | 5 | 13 | 0
Infusion Related Reaction (General disorders) | 13 | 0 | 0 | 0
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Gallbladder Pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anaphylaxis (Immune system disorders) | 1 | 0 | 0 | 0
Allergic Reaction (Immune system disorders) | 12 | 1 | 5 | 0
Infections And Infestations - Other (Infections and infestations) | 7 | 9 | 16 | 0
Wound Infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 8 | 19 | 9 | 0
Tooth Infection (Infections and infestations) | 4 | 0 | 0 | 0
Vulval Infection (Infections and infestations) | 1 | 0 | 1 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 0 | 1 | 0
Skin Infection (Infections and infestations) | 2 | 7 | 8 | 0
Sinusitis (Infections and infestations) | 5 | 6 | 7 | 0
Sepsis (Infections and infestations) | 3 | 3 | 2 | 0
Rhinitis Infective (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 2 | 0
Otitis Media (Infections and infestations) | 1 | 0 | 0 | 0
Papulopustular Rash (Infections and infestations) | 0 | 1 | 1 | 0
Nail Infection (Infections and infestations) | 0 | 0 | 0 | 1
Mucosal Infection (Infections and infestations) | 0 | 3 | 3 | 0
Lymph Gland Infection (Infections and infestations) | 0 | 1 | 0 | 0
Pelvic Infection (Infections and infestations) | 0 | 1 | 0 | 0
Lung Infection (Infections and infestations) | 2 | 4 | 5 | 1
Laryngitis (Infections and infestations) | 0 | 2 | 0 | 0
Kidney Infection (Infections and infestations) | 0 | 0 | 0 | 1
Eye Infection (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis Infective (Infections and infestations) | 0 | 0 | 1 | 0
Gum Infection (Infections and infestations) | 1 | 0 | 1 | 0
Vaginal Infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 19 | 25 | 38 | 0
Bronchial Infection (Infections and infestations) | 3 | 6 | 9 | 0
Enterocolitis Infectious (Infections and infestations) | 2 | 0 | 2 | 0
Bladder Infection (Infections and infestations) | 1 | 2 | 1 | 1
Lip Infection (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Injury, Poisoning And Procedural Complications - O (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Injury To Carotid Artery (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 7 | 5 | 0
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Burn (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 13 | 4 | 6 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Investigations - Other (Investigations) | 2 | 6 | 11 | 0
Weight Loss (Investigations) | 9 | 13 | 58 | 6
Weight Gain (Investigations) | 5 | 3 | 3 | 0
Serum Amylase Increased (Investigations) | 1 | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 67 | 21 | 40 | 4
Lymphocyte Count Decreased (Investigations) | 24 | 32 | 15 | 1
Lipase Increased (Investigations) | 0 | 0 | 1 | 0
Inr Increased (Investigations) | 3 | 1 | 4 | 0
Hemoglobin Increased (Investigations) | 0 | 0 | 4 | 0
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 0 | 1 | 0 | 0
Creatinine Increased (Investigations) | 12 | 41 | 33 | 1
Cholesterol High (Investigations) | 0 | 2 | 1 | 0
Neutrophil Count Decreased (Investigations) | 105 | 24 | 32 | 4
Urine Output Decreased (Investigations) | 0 | 1 | 0 | 0
Cardiac Troponin I Increased (Investigations) | 1 | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 4 | 6 | 11 | 0
White Blood Cell Decreased (Investigations) | 67 | 39 | 33 | 3
Aspartate Aminotransferase Increased (Investigations) | 17 | 9 | 18 | 5
Alkaline Phosphatase Increased (Investigations) | 14 | 8 | 17 | 3
Alanine Aminotransferase Increased (Investigations) | 14 | 9 | 21 | 5
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1 | 2 | 0
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 1 | 3 | 5 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0 | 5 | 0
Hyponatremia (Metabolism and nutrition disorders) | 16 | 26 | 31 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 32 | 7 | 22 | 0
Hypokalemia (Metabolism and nutrition disorders) | 24 | 15 | 31 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0 | 8 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 27 | 8 | 16 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 | 16 | 26 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypernatremia (Metabolism and nutrition disorders) | 4 | 2 | 5 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 6 | 5 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 22 | 40 | 25 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 3 | 6 | 0
Dehydration (Metabolism and nutrition disorders) | 12 | 15 | 20 | 0
Anorexia (Metabolism and nutrition disorders) | 37 | 52 | 78 | 9
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 18 | 27 | 29 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 21 | 23 | 0
Musculoskeletal Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 4 | 4 | 4 | 0
Muscle Weakness Left-Sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint Range Of Motion Decreased Lumbar Spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 14 | 10 | 25 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 6 | 3 | 1
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 13 | 7 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 22 | 34 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 23 | 22 | 0
Musculoskeletal And Connective Tissue Disorder - O (Musculoskeletal and connective tissue disorders) | 2 | 2 | 10 | 0
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 5 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Leukemia Secondary To Oncology Chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Nervous System Disorders - Other (Nervous system disorders) | 1 | 2 | 2 | 0
Trigeminal Nerve Disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 4 | 3 | 5 | 0
Transient Ischemic Attacks (Nervous system disorders) | 1 | 0 | 0 | 0
Stroke (Nervous system disorders) | 1 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 1 | 2 | 1 | 1
Seizure (Nervous system disorders) | 1 | 1 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 3 | 2 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 56 | 30 | 26 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 5 | 2 | 0 | 0
Paresthesia (Nervous system disorders) | 5 | 4 | 5 | 0
Neuralgia (Nervous system disorders) | 1 | 2 | 0 | 0
Memory Impairment (Nervous system disorders) | 5 | 3 | 5 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 2 | 0
Intracranial Hemorrhage (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 34 | 33 | 63 | 5
Extrapyramidal Disorder (Nervous system disorders) | 0 | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 9 | 25 | 30 | 2
Sinus Pain (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 4 | 1 | 0
Dizziness (Nervous system disorders) | 22 | 31 | 40 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Concentration Impairment (Nervous system disorders) | 2 | 0 | 0 | 0
Cognitive Disturbance (Nervous system disorders) | 1 | 3 | 5 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1 | 0
Psychiatric Disorders - Other (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Personality Change (Psychiatric disorders) | 0 | 1 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Libido Decreased (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 21 | 23 | 14 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 16 | 16 | 17 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 7 | 1 | 6 | 0
Anxiety (Psychiatric disorders) | 8 | 13 | 17 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1 | 0
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 2 | 5 | 6 | 0
Urinary Urgency (Renal and urinary disorders) | 10 | 5 | 2 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 5 | 4 | 4 | 0
Urinary Tract Pain (Renal and urinary disorders) | 4 | 11 | 7 | 0
Urinary Frequency (Renal and urinary disorders) | 5 | 9 | 8 | 0
Proteinuria (Renal and urinary disorders) | 4 | 11 | 17 | 4
Hematuria (Renal and urinary disorders) | 3 | 7 | 6 | 0
Cystitis Noninfective (Renal and urinary disorders) | 2 | 2 | 1 | 2
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 6 | 6 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 5 | 4 | 1
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Vaginal Pain (Reproductive system and breast disorders) | 1 | 2 | 3 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 3 | 5 | 2 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Perineal Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 3 | 3 | 4 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 3 | 4 | 1 | 0
Vaginal Inflammation (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 2 | 1 | 0
Breast Pain (Reproductive system and breast disorders) | 2 | 2 | 1 | 0
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 0
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 22 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 17 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 6 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 6 | 0
Pharyngeal Mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 15 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 26 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 6 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 | 45 | 52 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 35 | 44 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 6 | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 7 | 13 | 15 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 | 1 | 1 | 1
Scalp Pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 10 | 5 | 8 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 11 | 11 | 1
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 11 | 1 | 12 | 4
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 19 | 14 | 23 | 0
Nail Ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Nail Loss (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 9 | 2 | 14 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 14 | 20 | 1
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 0 | 0 | 1 | 0
Vascular Disorders - Other (Vascular disorders) | 0 | 1 | 0 | 0
Visceral Arterial Ischemia (Vascular disorders) | 0 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0
Thromboembolic Event (Vascular disorders) | 7 | 6 | 14 | 0
Superficial Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral Ischemia (Vascular disorders) | 0 | 0 | 1 | 0
Lymphedema (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 5 | 8 | 19 | 0
Hypertension (Vascular disorders) | 15 | 24 | 128 | 11
Hot Flashes (Vascular disorders) | 12 | 10 | 8 | 0
Flushing (Vascular disorders) | 4 | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT02446600/Prot_SAP_000.pdf